CLINICAL TRIAL: NCT06082622
Title: Evaluation of the Triple Management Program in the Management of Functional Chronic Constipation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Ahmed ElSayed A. Moustafa, Assistant professor of pediatric surgery, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: minia school of medicine
Record Dates: First submitted 2023-10-01; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Constipation Chronic Idiopathic
Keywords: constipation; pediatrics; ACE; non surgical
MeSH Terms: conditions — Constipation | interventions — Laxatives

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEW PROTOCOL (Experimental): Using the triple therapy protocol for management of FC
  Interventions: Combination Product: laxatives
- CONVENTIONAL (Experimental): Using the conventional laxative therapy with rehabilitation (two axis) only
  Interventions: Combination Product: laxatives

INTERVENTIONS:
Combination Product: laxatives — triple therapy of drugs, behaviour and mental axis

SUMMARY:
Abstract Background: Chronic constipation is a common disease in children, 3% all children visit gastroenterology clinics with different types and complains. It is very harsh, time consuming and psychological problems to a child and all his family members.

Objective: To find a simple and effective training method that manages the bowel habits intervals both easy and effective for both child and parents.

Patients and methods: A training program for 18 weeks in 180 children with follow up every three months for 3 years between March 2016 and April 2019. Two groups were assembled, Group (A) with 90 children managed by the 3 Role program and Group (B) formed of the other 90 children treated with traditional guidelines. All types of functional Constipations and all ages are distributed equally in the two Groups. The Parents were taught to Hang a Sign Saying (One Bowel habit by third day at least) and then follow the Triple method program for 18 weeks. First follow up is on the 3rd week. The triple axis program is working on mental, colon elasticity and fecal consistency. The Mental axis is done by bowel interval sets in fixed 3 times for 10 minutes in each, Colon contents by certain diet protocol and colon motility and elasticity by drugs.

DETAILED DESCRIPTION:
* Introduction Functional constipation (FC) is a common problem in children, with an estimated worldwide incidence of 9.5% . If there is no underlying organic reason, which is the case in up to 95% of children, constipation is classified as FC. The etiology of the 5% of cases with an organic origin range from metabolic to endocrine problems to Hirschsprung disease, anorectal malformations, and neuromuscular diseases. To diagnose Constipation in a child clinically, it is currently based on the pediatric diagnostic Rome IV criteria, Figure 1. Constipation poses a significant burden on both children and their family and is associated with a reduced quality of life, diminished academic performances and psychological problems including aggression, anxiety, depression, and altered emotional reactivity. Moreover, constipation is common in children with behavioral disorders, such as attention deficit hyperactivity disorder and autism spectrum disorders . Symptoms of FC may persist into adulthood despite adequate laxative treatment. The pathophysiology of constipation is multifactorial and incompletely understood. In more than 90 % of the cases, there is no organic explanation for the symptoms. Genetic predisposition, low-socio economic status, inadequate daily fiber intake, insufficient fluid intake, and immobility have been proposed as factors leading to FC. The most encountered etiological factor in children is withholding behavior, usually occurring after experiencing a painful or frightening evacuation of stools. Rome III criteria are commonly used to define functional constipation. Children with developmental age of at least 4 years must fulfill two or more of the following criteria. They should have insufficient criteria for diagnosis of irritable bowel syndrome. The criteria must be fulfilled at least once per week for at least 2 months before diagnosis. There should be no evidence of an organic disease explaining the symptoms .

  1. Two or fewer defecations in the toilet per week.
  2. At least one episode of fecal incontinence per week.
  3. History of retentive posturing or excessive volitional stool retention.
  4. History of painful or hard bowel movements.
  5. Presence of a large fecal mass in the rectum.
  6. History of large diameter stools. Almost identical criteria have been defined for infants and toddlers. Those criteria should be fulfilled for at least 1 month .
* Treatment regimens Conventional treatment of children with Functional Constipation involves non-pharmacological interventions (education, toilet training, defecation diary, and reward system) in combination with pharmacological interventions such as oral laxatives, of which poly-ethylene glycol is the first-line drug of choice.

Alternative treatment options for children with intractable constipation are limited and include anal sphincter botulinum toxin injections, trans anal irrigation, antegrade continent enemas (ACE), and, in rare cases, sacral nerve stimulation (SNS) and partial or total surgical resection of the colon15. and is frequently associated with fecal incontinence. In pediatrics, fecal incontinence has been defined as the voluntary or involuntary passage of feces into the underwear or in socially inappropriate places, in a child with a developmental age of at least 4 years. It has been suggested that in otherwise healthy children, fecal incontinence is secondary to 'overflow', and therefore results from the presence of constipation . This review aims to find a simple and effective training method that manages the bowel habits intervals both easy and effective for both child and parents. The exact prevalence of functional fecal incontinence associated with stool retention varies.

• Methodology A training program for 18 weeks in 180 children with follow up every three months for 3 years between March 2016 and April 2019. Two groups were assembled, Group (A) formed of the other 90 children treated with the 3 role program and Group (B) with 90 children managed by the previously mentioned traditional guidelines. All types of Constipations and all ages are distributed equally in the two Groups. The Parents in Group A were thought to Hang a Sign of (One Bowel habit by third day at least) and then follow the triple method program for 3 months. First follow up is on the 3rd week. The triple axis program is working on Psychic and mental axis, colon to retain its elasticity and fecal consistency.

I. The Mental axis (Gut-Brain interaction)

1. Habit timing training:

   It is done by bowel interval sets in fixed 3 times for 10-15 minutes of each, the preferred timing for training is just after breakfast, lunch and one hour before bedtime. The training is done to seek the regain of brain-Colon reflex and to bypass the psychic trauma of the child due to constipation with overflow which was wrongly diagnosed as incontinence. While the child was sitting in the toilet, no commands were directed to him/her. As there is no need to give a burden to his rehabilitation and to ensure that the axis is involuntarily done.

   Child is asked to leave the toilet even if there is no desire for defecation.
2. Exercise and daily activity:

   Increased daily activity and frequent exercise is favored to increase bowel movement and decrease psychic distress. Regular sports by fixed timing triple a week is encouraged.
3. Psychic therapy:

Family support is a golden axis for management progress, the feeling of security and backing plays an important role in fixing the problem and increase morale. Sometimes a child may need a psychiatric visit if it was a long time of constipation, and the overflow left a psychic trauma to the child.

II. The Pharmacological Colon Support That was done by trying to reduce the impacted colon load as to regain the lost or altered elasticity through the longtime of constipation and reabsorption of fluids through increased contact time between fecal matter and Intestine. The golden role that was informed to parents is that the hanged sign should be joined with drug protocol according to bowel evacuation intervals. So, another sign is drawn to parents with medication role related to bowel habits, to be easy remembered a card was designed as traffic light with Stop, Care and Go orders according to defecation modes Fig (2,3). An osmotic laxative medication (Lactulose) is thought to be a green light medication for a three-month period of program. If more than 24 hours with no defecation happened a yellow sign is hanged and a Na picosulphate drops is prescribed for the second day, if still no acceptable defecation retained, a red sign on the third day is waved and a local Enema with Mono/disodium phosphate is applied, then a green sign is regained. This regimen is maintained for three months and first follow-up with complete data on using the yellow or red sign is achieved within the first three weeks.

* Diet protocol As done with medication protocol, another traffic light card with instructions of which food can go (Green) as vegetables, Laxative fruits, and plenty of fluids. Other diet groups may be taken with caution (yellow) as Proteins, dairy products and low to medium doses of carbohydrates. While the last group (Red) should be quietly banned as conservatives contained diets, fats or constipating or citrus fruits. child is advised to take his main meals at a fixed time.
* Follow up. A Statistical sheet is delivered to parents to fulfill the numbers of bowel habits per day, how many times we had to take Picosulphate drops and/or Enemas? how many times has the child had soiled underwear? and how many times he succeeded in defecating during toilet training.

Figure 1: Rome IV disorders of chronic constipation5.

Child/Adolescent, 12

A minimum of 1 month of two or more of the following occurring at least once per week, with insufficient criteria for a diagnosis of irritable bowel:

* Two or fewer defecation in the toilet per week in a child of developmental age of at least 4 years.
* At least one episode of fecal incontinence per week.
* History of retentive posturing or excessive volitional stool retention.
* History of painful or hard bowel movements.
* Presence of a large fecal mass in the rectum.
* History of large diameter stools that can obstruct the toilet after appropriate evaluation, the symptoms cannot be fully explained by another medical condition.

After appropriate evaluation, the symptoms cannot be fully explained by another medical condition.

Figure 2: Traffic sign card of diet regimen.

Figure 3: Traffic sign card of drug protocol

One Bowel habit by third day at least.

Figure 4: The golden role sign.

ELIGIBILITY:
Inclusion Criteria:

* All types of Constipations and all ages are distributed equally in the two Groups

Exclusion Criteria:

* surgically treated

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
number of toilets per day | 3 days
  how many times the patient evacuate colon contents

IPD SHARING:
Plan to Share IPD: Yes
all eligible data to be shared will be available for researchers with organization domain addresses
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after manuscript is accepted to be published and it will be affordable for as long as it required
Access Criteria: by e-mail